CLINICAL TRIAL: NCT04938622
Title: Bioenergetics of Exercise-Induced Menstrual Disturbances
Acronym: BioE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Nancy Williams, Professor and Head, Department of Kinesiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 990878; R01HD039245-01 (NIH)
Record Dates: First submitted 2021-06-01; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Menstruation Disturbances; Luteal Phase Defect; Amenorrhea; Oligomenorrhea
Keywords: Energy Balance; Menstrual Cycle Disturbance; Luteal Phase Defect; Amenorrhea; Oligomenorrhea
MeSH Terms: conditions — Menstruation Disturbances; Amenorrhea; Oligomenorrhea | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sedentary Control (Experimental): Participants did not exercise but consumed a diet that has an appropriate number of calories to maintain body weight throughout the intervention (3 menstrual cycles).
  Interventions: Other: Sedentary Control
- Exercising control (Experimental): Participants exercised but were given extra calories to remain in energy balance throughout the intervention (3 menstrual cycles).
  Interventions: Other: Exercising control
- 15 percent energy deficit (ED1) (Experimental): Participants exercised for the equivalent of 15 percent of their daily caloric intake needs throughout the intervention cycles.
  Interventions: Other: 15 percent energy deficit
- 30 percent energy deficit (ED2) (Experimental): Participants exercised for the equivalent of 30 percent of their daily caloric intake needs throughout the intervention cycles.
  Interventions: Other: 30 percent energy deficit
- 30 percent energy deficit 15/15 (ED2) (Experimental): Participants exercised for the equivalent of 15 percent of their daily caloric intake needs throughout the intervention cycles, and their dietary intake was decreased by 15 percent to total a 30 percent energy deficit.
  Interventions: Other: 30 percent energy deficit (15/15)
- 60 percent energy deficit (ED3) (Experimental): Participants exercised for the equivalent of 30 percent of their daily caloric intake needs throughout the intervention cycles, and their dietary intake was decreased by 30 percent to total a 60 percent energy deficit.
  Interventions: Other: 60 percent energy deficit

INTERVENTIONS:
Other: Sedentary Control — Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had calories sufficient to maintain body weight. Diet composition was 55 percent carbohydrates, 30 percent fat, and 15 percent protein.
  Other Names: Diet
  Arms: Sedentary Control
Other: Exercising control — Exercise: Participants engaged in supervised exercise training in Noll Laboratory Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had calories sufficient to maintain body weight and additional calories to remain in energy balance. Diet composition was 55 percent carbohydrates, 30 percent fat, and 15 percent protein.
  Other Names: Diet
  Arms: Exercising control
Other: 15 percent energy deficit — Exercise: Participants engaged in supervised exercise training in Noll Laboratory that was equal to 15 percent of the participants' daily caloric needs.
  Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had calories to meet metabolic needs (before 15 percent deficit exercise). Diet composition was 55 percent carbohydrates, 30 percent fat, and 15 percent protein.
  Other Names: Diet and exercise
  Arms: 15 percent energy deficit (ED1)
Other: 30 percent energy deficit — Exercise: Participants engaged in supervised exercise training in Noll Laboratory that was equal to 30 percent of the participants' daily caloric needs.
  Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had calories to meet metabolic needs (before 30 percent deficit exercise). Diet composition was 55 percent carbohydrates, 30 percent fat, and 15 percent protein.
  Other Names: Diet and exercise
  Arms: 30 percent energy deficit (ED2)
Other: 30 percent energy deficit (15/15) — Exercise: Participants engaged in supervised exercise training in Noll Laboratory that was equal to 15 percent of the participants' daily caloric needs.
  Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had 15 percent less calories than those needed to meet metabolic needs. Diet composition was 55 percent carbohydrates, 30 percent fat, and 15 percent protein.
  Other Names: Diet and exercise
  Arms: 30 percent energy deficit 15/15 (ED2)
Other: 60 percent energy deficit — Exercise: Participants engaged in supervised exercise training in Noll Laboratory that was equal to 30 percent of the participants' daily caloric needs.
  Diet: Participants consumed meals in the General Clinical Research Center metabolic kitchen that had 30 percent less calories than those needed to meet metabolic needs. Diet composition was 55 percent carbohydrates, 30 percent fat, and 15 percent protein.
  Other Names: Diet and exercise
  Arms: 60 percent energy deficit (ED3)

SUMMARY:
Menstrual disturbances are frequently observed in physically active women and female athletes. Short term prospective studies have shown that diet and exercise interventions can lead to decreases in Luteinizing hormone (LH) pulsatility, however these studies are unable to capture further changes in menstrual status. One longer term prospective study over two menstrual cycles showed that weight loss elicited menstrual disturbances, but there were no quantifiable measurements of energy availability. Thus, the primary purpose of this study was to assess how varying levels of energy deficiency created through a combination of caloric restriction and exercise affect menstrual function in young, premenopausal, sedentary women.

DETAILED DESCRIPTION:
Long term energy deficiency in women can lead to functional hypothalamic amenorrhea (FHA), which can cause many health detriments such as osteopenia, stress fractures, transient infertility, dyslipidemia, and impaired endothelial function. Though studies involving diet and exercise interventions have shown how energy deficiency can lead to menstrual disturbances prospectively, this study aims to extend those findings by measuring the magnitude of energy deficit that could lead to these disturbances. Hypotheses for this study are: 1) there would be a dose-response relation between the induction of menstrual disturbances (luteal phase defects, anovulation, and oligomenorrhea) and the magnitude of energy deficiency such that the intervention groups experiencing a greater energy deficit would incur a significantly greater incidence of menstrual cycle disturbances and 2) the intervention groups experiencing a greater energy deficit would incur a greater incidence of more severe menstrual cycle disturbances.

The study included one baseline menstrual cycle and 3 intervention menstrual cycles. During the baseline period, participants were randomly assigned to an experimental group for intervention menstrual cycles 1, 2, and 3 of the study. The goal of the subject groupings was to test the impact of varying levels of an energy deficit created by the combination of caloric restriction and exercise on menstrual function. They were assigned to either a control group that did not exercise and consumed a number of calories estimated to maintain body weight, a control group that exercised but received extra food calories to remain in energy balance (EXCON), or one of four groups that exercised and were prescribed reduced energy intake to create varying levels of an energy deficit. Specifically, the four groups of energy deficit were 1) an increase of 15 percent kcal of exercise (15 percent deficit, ED1), 2) an increase of 30 percent kcal of exercise (30 percent deficit, ED2), 3) a decrease of 15 percent in dietary intake combined with an increase of 15 percent of exercise, (30 percent deficit 15/15, ED2), and 4) a decrease of 30 percent in dietary intake combined with an increase of 30 percent kcal of exercise (60 percent deficit, ED3). The number of participants for analysis was 34 participants in the following groups: EXCON (n = 8), ED1 (n = 6), ED2 (n = 12), and ED3 (n = 8).

Baseline energy needs were assessed during the baseline cycle. Resting metabolic rate and nonexercise physical activity were added to determine a caloric need for the day. Caloric intake was supervised throughout the entire study, and meals were comprised of 55 percent carbohydrates, 30 percent fat, and 15 percent protein. Exercise training was also supervised, and maximal oxygen consumption (VO2 max) was calculated. Menstrual status was assessed through analysis of daily urinary metabolites of estrone-1-glucuronide (E1G), pregnanediol glucuronide (PdG), and midcycle LH. Underwater weighing and a digital scale were used to assess body composition, and fasting blood samples were collected to assess metabolic hormones.

ELIGIBILITY:
Inclusion Criteria:

* Weight 45-75 kg
* Body fat 15-35 percent
* BMI 18-25 kg/m2
* Nonsmoking
* <1 hour/week of purposeful aerobic exercise for the past 6 months
* Documentation of at least two ovulatory menstrual cycles during screening.

Exclusion Criteria:

* History of serious medical conditions
* Medication use that would alter metabolic hormone levels
* Significant weight loss/gain (±2.3 kg) in the last year
* Current evidence of disordered eating or history of an eating disorder
* Taking exogenous hormonal contraceptives for the past 6 months

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2001-05-01 (Actual); Primary Completion 2005-04-30 (Actual); Study Completion 2005-04-30 (Actual)

PRIMARY OUTCOMES:
Change in frequency of menstrual disturbances (disturbances /cycle) | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC)
  Frequency of menstrual disturbances including luteal phase defects, anovulation, oligomenorrhea cycles, and anovulatory cycles analyzed by daily urinary metabolites of estrone-1-glucuronide (E1G), pregnanediol glucuronide (PdG), and midcycle LH

SECONDARY OUTCOMES:
Change in percent body fat | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC), & Post Study (days 1-7)
  Change in percent body fat (%)
Change in metabolic hormones | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, Mid- study (week 3 of MC during intervention MC 2) an (28 days (d) or the length of 1 MC), & Post Study (Days (d)1-7 of cycle
  Change in metabolic hormones total triiodothyronine (T3 ng/dL)) and insulin-like growth factor-1 (IGF-1 ng/ml).
Change in cycle length (days (d)) | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC)
  Change in cycle length (days (d))
Change in aerobic capacity | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, & Post Study (Days (d)1-7 of cycle
  Change in aerobic capacity, VO2 max (ml/kg/min)
Change in body weight | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC), & Post Study (days 1-7)
  Body weight (kg)
Change in fat mass | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC), & Post Study (days 1-7)
  Change in fat mass (kg)
Change in fat free mass | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC), & Post Study (days 1-7)
  Change in fat free mass (kg)
Change in follicular phase length | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC)
  Change in follicular phase length (days (d))
Change in luteal phase length | Baseline Menstrual Cycle (MC) (28 days (d) or the length of 1 MC, intervention MC 1 (28 days or the length of 1 MC), intervention MC 2 (28 days or the length of 1 MC), and intervention MC 3 (28 days or the length of 1 MC)
  Change in luteal phase length (days (d))

CONTACTS AND LOCATIONS:
Overall Officials: Nancy I Williams, ScD, Principal Investigator — Penn State University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lieberman JL, DE Souza MJ, Wagstaff DA, Williams NI. Menstrual Disruption with Exercise Is Not Linked to an Energy Availability Threshold. Med Sci Sports Exerc. 2018 Mar;50(3):551-561. doi: 10.1249/MSS.0000000000001451. PMID 29023359
- [Result] Williams NI, Leidy HJ, Hill BR, Lieberman JL, Legro RS, De Souza MJ. Magnitude of daily energy deficit predicts frequency but not severity of menstrual disturbances associated with exercise and caloric restriction. Am J Physiol Endocrinol Metab. 2015 Jan 1;308(1):E29-39. doi: 10.1152/ajpendo.00386.2013. Epub 2014 Oct 28. PMID 25352438